CLINICAL TRIAL: NCT02862080
Title: Impact of Combining tsDCS and Robotic Exoskeleton Gait Training on Spinal Excitability and Gait Function in Individuals With SCI
Brief Title: Combining tsDCS and Exoskeleton Gait Training on Spinal Excitability in SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: TIRR Memorial Hermann (Other)
Responsible Party: Principal Investigator, Marcie Kern, Research Physical Therapist, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0329
Record Dates: First submitted 2016-06-10; First posted 2016-08-10 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- no intervention; then no intervention; then cathode tsDCS + Ekso; then Ekso; then cathode tsDCS+Ekso (Experimental): Non-invasive transcutaneous spinal direct current stimulation (tsDCS) applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  Cathode tsDCS + Ekso will combine the use of cathode tsDCS application followed by a walking session in Ekso. Ekso will consist of a walking session in Ekso with no tsDCS.
  Interventions: Device: cathode tsDCS; Device: Ekso
- no intervention; then no intervention; then Ekso; then cathode tsDCS + Ekso; then Ekso (Experimental): Non-invasive transcutaneous spinal direct current stimulation (tsDCS) applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  Cathode tsDCS + Ekso will combine the use of cathode tsDCS application followed by a walking session in Ekso. Ekso will consist of a walking session in Ekso with no tsDCS.
  Interventions: Device: cathode tsDCS; Device: Ekso
- no intervention; then no intervention; then anode tsDCS + Ekso; then Ekso; then anode tsDCS + Ekso (Experimental): Non-invasive transcutaneous spinal direct current stimulation (tsDCS) applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  Anode tsDCS + Ekso will combine the use of anode tsDCS application followed by a walking session in Ekso. Ekso will consist of a walking session in Ekso with no tsDCS.
  Interventions: Device: Ekso; Device: anode tsDCS
- no intervention; then no intervention; then Ekso; then anode tsDCS + Ekso; then Ekso (Experimental): Non-invasive transcutaneous spinal direct current stimulation (tsDCS) applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  Anode tsDCS + Ekso will combine the use of anode tsDCS application followed by a walking session in Ekso. Ekso will consist of a walking session in Ekso with no tsDCS.
  Interventions: Device: Ekso; Device: anode tsDCS

INTERVENTIONS:
Device: cathode tsDCS — Non-invasive electrical stimulation, transcutaneous spinal direct current stimulation (tsDCS) is the application of electrical current to the spinal cord via surface electrodes placed on the skin.
  Arms: no intervention; then no intervention; then Ekso; then cathode tsDCS + Ekso; then Ekso; no intervention; then no intervention; then cathode tsDCS + Ekso; then Ekso; then cathode tsDCS+Ekso
Device: Ekso — Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
Device: anode tsDCS — Non-invasive electrical stimulation, transcutaneous spinal direct current stimulation (tsDCS) is the application of electrical current to the spinal cord via surface electrodes placed on the skin.
  Arms: no intervention; then no intervention; then Ekso; then anode tsDCS + Ekso; then Ekso; no intervention; then no intervention; then anode tsDCS + Ekso; then Ekso; then anode tsDCS + Ekso

SUMMARY:
The purpose of the study is to determine whether transcutaneous spinal direct current stimulation (tsDCS) is safe for individuals with spinal cord injury (SCI). tsDCS is an electrical current applied to the skin. The plan is to also study the potential neurophysiological changes (changes in speed and excitability of the nerves) and functional improvements in gait (for example, gait quality, speed and walking distance) for individuals with SCI after combined application of tsDCS and exoskeleton assisted gait training.

DETAILED DESCRIPTION:
Subjects will participate in two baseline visits, 4 days apart. Each baseline visit will last 1 hour and will include assessment of soleus H-Reflex and 10 meter walk test on arrival and 40 minutes after the initial assessment. Subjects will be asked to minimize their activity between assessments by either sitting in a chair or lying on a mat.

Each training visit will involve either an exoskeleton intervention or a combined exoskeleton and tsDCS intervention. Each training visit will include assessment of soleus H-Reflex and 10 meter walk test before and after the exoskeleton intervention or before and after the combined exoskeleton and tsDCS intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female
* ≥18 years of age
* Able to achieve adequate fit within exoskeleton
* Diagnosis of spinal cord injury (SCI), T10 level and above (T11 and 12 may participate if no clinical signs of lower motor neuron lesion present)
* Minimum of 6 months post injury
* Sufficient range of motion to attain normal, reciprocal gait pattern, and transition from normal sit to stand or stand to sit
* Weight <220 pounds
* Intact skin on all surfaces in contact with device and load bearing surfaces
* Ability to perform informed consent

Exclusion Criteria:

* Pregnancy
* Spinal instability
* Unhealed limb or pelvic fractures or any condition restricting weight bearing in limbs
* Presence of peripheral neuropathy or any pathology that could influence reflex excitability
* Diagnosis of other neurological injury other than SCI such as stroke/cerebrovascular accident (CVA), multiple sclerosis (MS), acquired brain injury (ABI), cerebral palsy (CP)
* Uncontrolled spasticity (≥3 on Modified Ashworth Scale)
* Colostomy
* Decreased range of motion or contractures in legs (>10° at hips, knees or ankles)
* Uncontrolled autonomic dysreflexia
* Unresolved deep vein thrombosis
* Inability to tolerate standing due to cardiovascular issues or orthostatic hypotension
* Severe comorbidities: active infections, heart, lung, or circulatory conditions
* Pressure sores, impaired skin integrity
* Use of mechanical ventilation for respiratory support
* Presence of any of the following contraindications to electrical stimulation: cardiac pacemaker, deep brain stimulator, or evidence of cancerous (malignant) tissue
* Presence of metal in thoracic spine or region of electrode placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcie Kern, PT, MSPT, Principal Investigator — TIRR Memorial Hermann
Locations (1):
- NeuroRecovery Research Center at TIRR Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- no Intervention; Then no Intervention; Then Cathode tsDCS + Ekso; Then Ekso; Then Cathode tsDCS+Ekso; no Intervention; Then no Intervention; Then Ekso; Then Cathode tsDCS + Ekso; Then Ekso: Non-invasive transcutaneous spinal direct current stimulation (tsDCS) applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  Cathode tsDCS + Ekso will combine the use of cathode tsDCS application followed by a walking session in Ekso. Ekso will consist of a walking session in Ekso with no tsDCS.
  cathode tsDCS: Non-invasive electrical stimulation, transcutaneous spinal direct current stimulation (tsDCS) is the application of electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso: Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
- no Intervention; Then no Intervention; Then Anode tsDCS + Ekso; Then Ekso; Then Anode tsDCS + Ekso; no Intervention; Then no Intervention; Then Ekso; Then Anode tsDCS + Ekso; Then Ekso: Non-invasive transcutaneous spinal direct current stimulation (tsDCS) applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  Anode tsDCS + Ekso will combine the use of anode tsDCS application followed by a walking session in Ekso. Ekso will consist of a walking session in Ekso with no tsDCS.
  Ekso: Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  anode tsDCS: Non-invasive electrical stimulation, transcutaneous spinal direct current stimulation (tsDCS) is the application of electrical current to the spinal cord via surface electrodes placed on the skin.
Period: 7 Days Before Any Intervention
Arm/Group | no Intervention; Then no Intervention; Then Cathode tsDCS + Ekso; Then Ekso; Then Cathode tsDCS+Ekso | no Intervention; Then no Intervention; Then Ekso; Then Cathode tsDCS + Ekso; Then Ekso | no Intervention; Then no Intervention; Then Anode tsDCS + Ekso; Then Ekso; Then Anode tsDCS + Ekso | no Intervention; Then no Intervention; Then Ekso; Then Anode tsDCS + Ekso; Then Ekso
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: 3 Days Before Any Intervention
Arm/Group | no Intervention; Then no Intervention; Then Cathode tsDCS + Ekso; Then Ekso; Then Cathode tsDCS+Ekso | no Intervention; Then no Intervention; Then Ekso; Then Cathode tsDCS + Ekso; Then Ekso | no Intervention; Then no Intervention; Then Anode tsDCS + Ekso; Then Ekso; Then Anode tsDCS + Ekso | no Intervention; Then no Intervention; Then Ekso; Then Anode tsDCS + Ekso; Then Ekso
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 1 (1 Week)
Arm/Group | no Intervention; Then no Intervention; Then Cathode tsDCS + Ekso; Then Ekso; Then Cathode tsDCS+Ekso | no Intervention; Then no Intervention; Then Ekso; Then Cathode tsDCS + Ekso; Then Ekso | no Intervention; Then no Intervention; Then Anode tsDCS + Ekso; Then Ekso; Then Anode tsDCS + Ekso | no Intervention; Then no Intervention; Then Ekso; Then Anode tsDCS + Ekso; Then Ekso
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | no Intervention; Then no Intervention; Then Cathode tsDCS + Ekso; Then Ekso; Then Cathode tsDCS+Ekso | no Intervention; Then no Intervention; Then Ekso; Then Cathode tsDCS + Ekso; Then Ekso | no Intervention; Then no Intervention; Then Anode tsDCS + Ekso; Then Ekso; Then Anode tsDCS + Ekso | no Intervention; Then no Intervention; Then Ekso; Then Anode tsDCS + Ekso; Then Ekso
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 2 (1 Week)
Arm/Group | no Intervention; Then no Intervention; Then Cathode tsDCS + Ekso; Then Ekso; Then Cathode tsDCS+Ekso | no Intervention; Then no Intervention; Then Ekso; Then Cathode tsDCS + Ekso; Then Ekso | no Intervention; Then no Intervention; Then Anode tsDCS + Ekso; Then Ekso; Then Anode tsDCS + Ekso | no Intervention; Then no Intervention; Then Ekso; Then Anode tsDCS + Ekso; Then Ekso
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | no Intervention; Then no Intervention; Then Cathode tsDCS + Ekso; Then Ekso; Then Cathode tsDCS+Ekso | no Intervention; Then no Intervention; Then Ekso; Then Cathode tsDCS + Ekso; Then Ekso | no Intervention; Then no Intervention; Then Anode tsDCS + Ekso; Then Ekso; Then Anode tsDCS + Ekso | no Intervention; Then no Intervention; Then Ekso; Then Anode tsDCS + Ekso; Then Ekso
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 1 Again (1 Week)
Arm/Group | no Intervention; Then no Intervention; Then Cathode tsDCS + Ekso; Then Ekso; Then Cathode tsDCS+Ekso | no Intervention; Then no Intervention; Then Ekso; Then Cathode tsDCS + Ekso; Then Ekso | no Intervention; Then no Intervention; Then Anode tsDCS + Ekso; Then Ekso; Then Anode tsDCS + Ekso | no Intervention; Then no Intervention; Then Ekso; Then Anode tsDCS + Ekso; Then Ekso
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ekso Alone, and Ekso + Cathode tsDCS: Participants received Ekso alone and also Ekso combined with cathode non-invasive transcutaneous spinal direct current stimulation (tsDCS).
  Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  tDCS applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso alone will consist of a walking session in Ekso with no tsDCS. Cathode tsDCS plus Ekso involves cathode tsDCS application followed by a walking session in Ekso.
- Ekso Alone, and Ekso + Anode tsDCS: Participants received Ekso alone and also Ekso combined with anode non-invasive transcutaneous spinal direct current stimulation (tsDCS).
  Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  tDCS applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Ekso alone will consist of a walking session in Ekso with no tsDCS. Anode tsDCS plus Ekso involves anode tsDCS application followed by a walking session in Ekso.
- Total: Total of all reporting groups
Arm/Group | Ekso Alone, and Ekso + Cathode tsDCS | Ekso Alone, and Ekso + Anode tsDCS | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.7) | 37 (9.9) | 39.5 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4
Level of Spinal Cord Injury (SCI) [Count of Participants; unit: Participants] — The level of injury is based on International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI). The level reported is the lowest (most caudal) segment of the spinal cord that remains fully intact for sensory and motor function. C is cervical (the region of the neck), with C1 being the highest level closest to the skull and C7 being the bottom of the neck. T is the thoracic/chest region (all the levels with ribs attached), with T1 being the top closest to the neck and T12 the bottom close to low back.
  Participants
    T1 | 1 | 0 | 1
    T9 | 0 | 1 | 1
    C5 | 1 | 1 | 2
Time since injury [Mean (Standard Deviation); unit: years] | 16.5 (16.26) | 6 (1.41) | 11.25 (11.21)

OUTCOME MEASURES:

1. Primary Outcome: Change in Spinal Cord Excitability as Measured by Percent Change in Soleus H-Reflex From Beginning of Session to End of the Same Session
Description: This visit includes assessment of soleus H-Reflex on arrival and 40 minutes after the initial assessment--change between these two readings is reported. Subjects will be asked to minimize their activity between the two assessments by either sitting in a chair or lying on a mat.
  The H-reflex is a reaction of muscles after electrical stimulation (this stimulation is not the intervention, but is instead part of the H-reflex assessment). H-reflex will be elicited by placing the cathode of an electrical stimulator in the popliteal fossa (a shallow depression located at the back of the knee joint) and stimulating the tibial nerve. To record the electrical-induced muscle activity (that is, to measure H-reflexes), surface electromyography electrodes will be placed at the soleus muscle of the testing leg.
Time Frame: beginning and end of first no-intervention visit (7 days before any intervention)
Population: All participants were assessed for the H-Reflex at this visit.
Measure: Mean (Standard Deviation); unit: percent change in H-Reflex
Groups:
- No Intervention: Neither Ekso nor tsDCS are applied.
Arm/Group | No Intervention
Number analyzed (Participants) | 4
percent change in H-Reflex | -3.13 (18.27)

2. Primary Outcome: Change in Spinal Cord Excitability as Assessed by Percent Change in Soleus H-Reflex From Beginning of Session to End of the Same Session
Description: as for outcome 1
Time Frame: beginning and end of second no-intervention visit (3 days before any intervention)
Population: All participants were assessed for the H-Reflex at this visit.
Measure: Mean (Standard Deviation); unit: percent change in H-Reflex
Arm/Group | No Intervention
Number analyzed (Participants) | 4
percent change in H-Reflex | -5.74 (10.96)

3. Primary Outcome: Change in Spinal Cord Excitability as Assessed by Percent Change in Soleus H-Reflex From Beginning of Session to End of the Same Session
Description: Soleus H-Reflex is assessed on arrival and then after the intervention is applied--change between these two readings is reported.
  The H-reflex is a reaction of muscles after electrical stimulation (this stimulation is not the intervention, but is instead part of the H-reflex assessment). H-reflex will be elicited by placing the cathode of an electrical stimulator in the popliteal fossa (a shallow depression located at the back of the knee joint) and stimulating the tibial nerve. To record the electrical-induced muscle activity (that is, to measure H-reflexes), surface electromyography electrodes will be placed at the soleus muscle of the testing leg.
Time Frame: before and after intervention on day 1
Population: All participants received all interventions as assigned during all 3 intervention periods and were assessed for H-reflex. For the cathode tsDCS + Ekso arm, 1 received the intervention once, and 1 received the intervention twice (3 data points total). For the anode tsDCS + Ekso arm, 1 received the intervention once, and 1 received the intervention twice (3 data points total). For the Ekso alone arm, 2 received the intervention once, and 2 received the intervention twice (6 data points total).
Measure: Mean (Standard Deviation); unit: percent change in H-Reflex
Units Other Than Participants: data points
Groups:
- Cathode tsDCS + Ekso: Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  tsDCS applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Cathode tsDCS plus Ekso involves cathode tsDCS application followed by a walking session in Ekso.
- Anode tsDCS + Ekso: Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  tsDCS applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Anode tsDCS plus Ekso involves anode tsDCS application followed by a walking session in Ekso.
- Ekso Alone: Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  Ekso alone will consist of a walking session in Ekso with no tsDCS.
Arm/Group | Cathode tsDCS + Ekso | Anode tsDCS + Ekso | Ekso Alone
Number analyzed (Participants) | 2 | 2 | 4
Number analyzed (data points) | 3 | 3 | 6
percent change in H-Reflex | 4.52 (6.47) | 11.19 (37.94) | 2.71 (13.06)

4. Primary Outcome: Change in Spinal Cord Excitability as Assessed by Percent Change in Soleus H-Reflex From Beginning of Session to End of the Same Session
Description: as for outcome 3
Time Frame: before and after intervention on day 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change in H-Reflex
Units Other Than Participants: data points
Arm/Group | Cathode tsDCS + Ekso | Anode tsDCS + Ekso | Ekso Alone
Number analyzed (Participants) | 2 | 2 | 4
Number analyzed (data points) | 3 | 3 | 6
percent change in H-Reflex | -2.30 (2.65) | -7.44 (24.82) | -9.82 (9.73)

5. Secondary Outcome: Gait Speed as Assessed by 10 Meter Walk Test
Description: The 10 Meter Walk Test (10MWT) will assess subject's gait speed. Four marks will be placed on the ground at 0, 2, 12 and 14 meters. Subjects will walk a total of 14 meters. The middle 10 meters (between marks at 2 and 12 meters) will be timed and recorded as their gait speed.
Time Frame: first no-intervention visit (7 days before any intervention)
Population: All participants were assessed for the 10MWT at this visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Intervention
Number analyzed (Participants) | 4
seconds | 37.14 (20.25)

6. Secondary Outcome: Gait Speed as Assessed by 10 Meter Walk Test
Description: as for outcome 5
Time Frame: second no-intervention visit (3 days before any intervention)
Population: One participant was not assessed for gait speed at this visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Intervention
Number analyzed (Participants) | 3
seconds | 27.20 (12.20)

7. Secondary Outcome: Gait Speed as Assessed by 10 Meter Walk Test
Description: Subjects will undergo a walking session with Ekso, Ekso will then be removed, and subjects will then perform a 10 Meter Walk Test (10MWT) without use of Ekso exoskeleton. The 10MWT will assess subject's gait speed. Four marks will be placed on the ground at 0, 2, 12 and 14 meters. Subjects will walk a total of 14 meters. The middle 10 meters (between marks at 2 and 12 meters) will be timed and recorded as their gait speed.
Time Frame: Day 1 of intervention
Population: All participants received all interventions as assigned during all 3 intervention periods and were assessed for gait speed. For the cathode tsDCS + Ekso arm, 1 received the intervention once, and 1 received the intervention twice (3 data points total). For the anode tsDCS + Ekso arm, 1 received the intervention once, and 1 received the intervention twice (3 data points total). For the Ekso alone arm, 2 received the intervention once, and 2 received the intervention twice (6 data points total).
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: data points
Arm/Group | Cathode tsDCS + Ekso | Anode tsDCS + Ekso | Ekso Alone
Number analyzed (Participants) | 2 | 2 | 4
Number analyzed (data points) | 3 | 3 | 6
seconds | 38.37 (14.47) | 41.64 (21.34) | 30.47 (20.43)

8. Secondary Outcome: Gait Speed as Assessed by 10 Meter Walk Test
Description: as for outcome 7
Time Frame: Day 2 of intervention
Population: One participant was not assessed for gait speed for two intervention periods of the cathode tsDCS + Ekso arm and one intervention period of the the Ekso alone arm. For the cathode tsDCS + Ekso arm, 1 received the intervention once (1 data point total). For the anode tsDCS + Ekso arm, 1 received the intervention once, and 1 received the intervention twice (3 data points total). For the Ekso alone arm, 1 received the intervention once, and 2 received the intervention twice (5 data points total).
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: data points
Arm/Group | Cathode tsDCS + Ekso | Anode tsDCS + Ekso | Ekso Alone
Number analyzed (Participants) | 1 | 2 | 3
Number analyzed (data points) | 1 | 3 | 5
seconds | 24.28 (0) | 37.53 (17.18) | 24.21 (13.01)

9. Secondary Outcome: Gait Speed as Assessed by 10 Meter Walk Test
Description: as for outcome 7
Time Frame: Day 3 of intervention
Population: One participant was not assessed for gait speed for two intervention periods of the cathode tsDCS + Ekso arm and one period of the the Ekso alone arm. Another participant was not assessed for gait speed for one period of the the anode tsDCS+Ekso arm. For the cathode tsDCS+Ekso arm, 1 received intervention once (1 data point). For the anode tsDCS+Ekso arm, 2 received intervention once (2 data points). For the Ekso alone arm, 1 received intervention once, and 2 received it twice (5 data points).
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: data points
Arm/Group | Cathode tsDCS + Ekso | Anode tsDCS + Ekso | Ekso Alone
Number analyzed (Participants) | 1 | 2 | 3
Number analyzed (data points) | 1 | 2 | 5
seconds | 16.42 (0) | 26.85 (15.07) | 22.98 (9.62)

10. Secondary Outcome: Gait Speed as Assessed by 10 Meter Walk Test
Description: as for outcome 7
Time Frame: Day 4 of intervention
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: data points
Arm/Group | Cathode tsDCS + Ekso | Anode tsDCS + Ekso | Ekso Alone
Number analyzed (Participants) | 1 | 2 | 5
Number analyzed (data points) | 1 | 3 | 5
seconds | 17.79 (0) | 38.43 (19.06) | 21.92 (7.87)

11. Secondary Outcome: Gait Speed as Assessed by 10 Meter Walk Test
Description: as for outcome 7
Time Frame: Day 5 of intervention
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: data points
Arm/Group | Cathode tsDCS + Ekso | Anode tsDCS + Ekso | Ekso Alone
Number analyzed (Participants) | 2 | 2 | 4
Number analyzed (data points) | 3 | 3 | 6
seconds | 39.38 (17.82) | 35.35 (18.51) | 26.43 (12.93)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Cathode tsDCS + Ekso: Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  tDCS applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Cathode tsDCS plus Ekso involves cathode tsDCS application followed by a walking session in Ekso.
- Anode tsDCS + Ekso: Ekso is a type of wearable robotic exoskeleton that provides support to an individual with lower extremity paralysis for standing and walking.
  tDCS applies electrical current to the spinal cord via surface electrodes placed on the skin.
  Anode tsDCS plus Ekso involves anode tsDCS application followed by a walking session in Ekso.
Arm/Group | Cathode tsDCS + Ekso | Anode tsDCS + Ekso | Ekso Alone | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT02862080/Prot_SAP_000.pdf